CLINICAL TRIAL: NCT03817073
Title: Assessing Fatiguability of Tongue Muscles and the Effect on Tongue Strength and Swallowing Pressures in Patients With Multiple Sclerosis
Brief Title: Assessing Fatiguability of Tongue Muscles in MS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Thomas More Kempen (Other)
Collaborators: Revalidatie & MS Centrum Overpelt (Other)
Responsible Party: Principal Investigator, Jan Vanderwegen, Principal Investigator, Clinical Professor, Thomas More Kempen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: TMALA19JVDW01
Record Dates: First submitted 2019-01-08; First posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Muscle Weakness; Fatigue; Multiple Sclerosis; Deglutition Disorders; Exertion; Excess
MeSH Terms: conditions — Muscle Weakness; Fatigue; Multiple Sclerosis; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iowa Oral Performance Instrument (IOPI) (Experimental): All MS patients will be included in this arm to compare with a historical control arm. Iowa Oral Performance Instrument (IOPI).
  Interventions: Device: Iowa Oral Performance Instrument (IOPI)

INTERVENTIONS:
Device: Iowa Oral Performance Instrument (IOPI) — Using biofeedback to attain repetitions of 80% of baseline MIP.

SUMMARY:
Multiple Sclerosis (MS) patients with subjective dysphagia will be tested for tongue strength fatigue using a strictly defined fatigue paradigm. A maximum of 40 sets will be performed, each set consisting of 5 repetitions of 80% of maximum isometric pressure (MIP) at the anterior tongue, followed by a MIP at the anterior tongue. Cut-off criteria are a MIP <50% of the baseline MIP, pronounced subjective discomfort and/or exceeding the allocated test time of 30 minutes.

DETAILED DESCRIPTION:
Eligibility is Mini-Mental State Exam-score (MMSE) > 23, a Eating Assessment Tool-score (EAT-10) > 3, or a Functional Oral Intake Scale-score (FOIS) < 7, or failing the Yale Swallow Protocol.

ELIGIBILITY:
Inclusion Criteria:

* proven MS
* subjective dysphagia

Exclusion Criteria:

* MMSE < 23
* major head and neck surgery
* history of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of successful repetitions | 30 minutes
  The number of repetitions where the target force was developed.
Evolution of MIP during subsequent repetitions | 30 minutes
  The change in MIP after each 5 repetitions.

SECONDARY OUTCOMES:
Baseline MIP as predictor for number of repetitions | 30 minutes
  Does baseline MIP predict the number of successful repetitions.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vanderwegen, Principal Investigator — Thomas More University College
Locations (1):
- Thomas More University College of Applied Sciences, Antwerp, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: No